CLINICAL TRIAL: NCT02855541
Title: Health Effects of Increasing Muscle Activation While Sitting in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, James Peterman, Graduate Student, University of Colorado, Boulder
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UColoradoBoulder
Record Dates: First submitted 2016-07-29; First posted 2016-08-04 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Blood Pressure
Keywords: Blood Glucose; Physical Fitness; Body Composition; Lipids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cycling intervention (Experimental): Participants will use a small cycling device (DeskCycle) at their workstation for 15 minutes every hour that they are at work.
  Interventions: Device: DeskCycle

INTERVENTIONS:
Device: DeskCycle — A small cycling ergometer that can fit under a desk at the workplace.

SUMMARY:
Previous research suggests that prolonged sitting increases risk for cardiometabolic diseases and the risk factors associated with cardiometabolic diseases. However, no study to date has examined if a chronic intervention that breaks up prolonged sitting in a real-world environment results in a reduction in the metabolic risk factors associated with cardiometabolic diseases. Thus, the objective of this study is to examine the potential health benefits of breaking up sitting bouts throughout the workday using a small cycling device (DeskCycle) in office workers involved with jobs that require prolonged bouts of sitting. The investigators hypothesize that breaking up sitting will be associated with improvements in cardiometabolic disease risk factors. More specifically, the investigators hypothesize that breaking up sitting will decrease blood glucose during an oral glucose tolerance test (OGTT), increase cardiorespiratory fitness (VO2max), decrease blood pressure, decrease body fat, increase HDL cholesterol, and decrease LDL cholesterol, total cholesterol, and triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females
* Subjects will need to be 18-55 years old
* Subjects will need to be sitting at least 6 hours/day on 5 days/week
* Subjects will need to be exercising less than 5 hour/week

Exclusion Criteria:

* Females that are pregnant or breast-feeding.
* Subjects must be free from any acute or chronic physical condition that would influence the outcome measures of the protocol. Examples include, but are not limited to advanced chronic disease states (chronic kidney, liver, heart, or lung disease), morbid obesity, emphysema, and an inability to use the legs for normal locomotion. Normality will be established on the basis of clinical history, physical exam, and vital signs. Any subject with a history of an uncontrolled metabolic disorder/disease or symptoms of active illness will be excluded from study. Any subject with a history of an uncontrolled metabolic disorder/disease such as diabetes (Type I or Type II) or symptoms of active illness will be excluded from study.

  * Subjects will be excluded if they have a fasted blood glucose level >126 mg/dl or a systolic blood pressure >140 mmHg.
* Medical/psychiatric/sleep disorders history: any clinically significant unstable medical or psychological condition within the last year (treated or untreated).
* Drug use:

  * Use of any medications, including over-the-counter and herbal products, that may affect metabolic function within 1 month prior to the study or need to use any of these medications at any time during the study (self-report by interview). Examples of potential medications that will exclude a subject include: beta-adrenergic blockers, sulfonylureas, biguanides, thiazolidinediones, alpha-glucosidase inhibitors, meglitinides, and dipeptidyl peptidase IV inhibitors. Note, subjects may be tested at a later date.
  * Use of any investigational drug within 1 month before the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cycling Intervention
Started | 25
Completed | 21
Not Completed | 4
Not completed — Change in health status | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Maximum Oxygen Consumption (VO2max) [Mean (Standard Deviation); unit: L/min] | 2.07 (0.44)
Blood Glucose [Mean (Standard Deviation); unit: mmol/L] — 2-h Post Oral Glucose Tolerance Test Blood Glucose
  mmol/L | 5.41 (1.21)
Work Sitting [Mean (Standard Deviation); unit: hours] | 7.04 (0.78)
HDL Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.09 (0.17)
LDL Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 2.50 (0.67)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.16 (0.64)
Lean Mass [Mean (Standard Deviation); unit: kg] | 47.8 (8.1)
Fat Mass [Mean (Standard Deviation); unit: kg] | 28.5 (13.0)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 112.2 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose
Description: 2-h Post Oral Glucose Tolerance Test Blood Glucose
Time Frame: Measured after 4 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
mmol/L | 5.60 (1.23)

2. Primary Outcome: Maximum Oxygen Consumption
Description: Maximum oxygen consumption (VO2max) will be used to determine physical fitness
Time Frame: Measured after 4 weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
L/min | 2.17 (0.44)

3. Secondary Outcome: Systolic Blood Pressure
Time Frame: Measured after 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
mmHg | 110.9 (12.5)

4. Secondary Outcome: HDL Cholesterol
Time Frame: Measured after 4 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
mmol/L | 1.17 (0.24)

5. Secondary Outcome: LDL Cholesterol
Time Frame: Measured after 4 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
mmol/L | 2.60 (0.59)

6. Secondary Outcome: Triglycerides
Time Frame: Measured after 4 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
mmol/L | 1.17 (0.72)

7. Secondary Outcome: Lean Mass
Time Frame: Measured after 4 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
kg | 47.4 (8.3)

8. Secondary Outcome: Fat Mass
Time Frame: Measured after 4 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cycling Intervention
Number analyzed (Participants) | 21
kg | 28.1 (13.2)

ADVERSE EVENTS:
Time Frame: 2 years.
Description: All-cause mortality was not assessed/collected.
Arm/Group | Cycling Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Participants were encouraged to cycle a set amount but this may not reflect how they would prefer to use the cycling device. In addition, the intervention was only 4 weeks long and more time may be needed to see improvements in the outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT02855541/Prot_SAP_000.pdf